CLINICAL TRIAL: NCT02228967
Title: Feasibility and Pilot Testing of SBI to Reduce Alcohol Misuse Among Active Duty Members in a Military ER Setting
Brief Title: Alcohol Screening, Brief Intervention, and Referral to Treatment in a Military Treatment Facility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Collaborators: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Responsible Party: Principal Investigator, Mark Reed, PhD, Director, San Diego State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: W81XWH-14-2-0014; 12019006 (Other Grant/Funding Number: Congressionally Directed Medical Research Programs)
Record Dates: First submitted 2014-08-26; First posted 2014-08-29 (Estimated); Results first posted 2019-07-25 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-08

CONDITIONS: Alcohol Dependency
Keywords: Alcohol Use; SBIRT; Military; Health Behavior; Emergency Room; Health Promotion; Formative Research; Randomized Trial
MeSH Terms: conditions — Alcoholism; Alcohol Drinking; Health Behavior; Emergencies | interventions — Mass Screening; Crisis Intervention; Motivational Interviewing

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (No Intervention): Those participants assigned to the usual care control group will be given a brochure on safe drinking limits, will be reminded of the 6-month follow-up, and thanked for their time.
- SBIRT (Active Comparator): Those assigned to the SBIRT intervention group will receive 1 of 3 tracks:
  1. Brief Intervention (BI) for At Risk Individuals (scores lower than 15) - Brief motivational intervention with feedback related to their use and change strategies.
  2. Brief Treatment (BT) for High Risk Individuals (scores of 16-19) - Brief Intervention on site and be offered 6 individual confidential sessions with a civilian Brief Treatment Counselor over the phone.
  3. Referral to Treatment (RT) for Severe Risk Individuals (scores of 20-40) - Brief Intervention on site and will be given a list of services where they may self-refer for further assessment and support.
  Interventions: Behavioral: SBIRT

INTERVENTIONS:
Behavioral: SBIRT — SBIRT is an "opportunistic" approach whereby patients are screened by Health Educators for their alcohol use, and then, taking advantage of a "teachable moment," are delivered a brief, motivational intervention matched to their level of risk.
  Other Names: Screening; Brief Intervention; Brief Treatment; Referral to Treatment; Motivational Interviewing
  Arms: SBIRT

SUMMARY:
An alcohol Screening, Brief Intervention and Referral to Treatment (SBIRT) approach will be adapted for use in a large military hospital setting, and then pilot tested in a military emergency department (ED) to assess its potential for effectiveness and for further testing in a large-scale trial. SBIRT is an "opportunistic" approach whereby all adult patients in the ED are screened by Health Educators for their alcohol use, and then, taking advantage of a "teachable moment," are delivered a brief, motivational intervention matched to their level of risk.

The feasibility/formative research activities in the first phase (Phase I) of the study are not summative research, and therefore, do not lend themselves to testable hypotheses. Hypotheses with regard to the pilot randomized trial in Phase II are as follows:

1. Participants in the SBIRT intervention will show relatively greater reductions over a six month period (or less increase) than the brochure/usual care control group in the prevalence of past-month heavy drinking, frequency of heavy drinking, past week number of drinks, and the AUDIT-based drinkers' index.
2. Alcohol use-related motivation/readiness to change and controlled drinking self-efficacy will show greater change in the SBIRT intervention group relative to the brochure/usual care control group.

   In addition, exploratory analyses will examine the following:
3. Sociodemographic/military variables (e.g., age, race/ethnicity, gender, branch of service, officer/enlisted status, PTS) and social-psychological factors (e.g., baseline readiness to change, self efficacy) will mediate or moderate changes in alcohol misuse.

DETAILED DESCRIPTION:
Deployment frequency and duration and combat exposure are implicated as risk factors for alcohol misuse and PTSD among military personnel. During the past 10 years, Department of Defense healthcare systems have observed steep increases in mental health and substance use services among personnel demobilizing from these conflicts. Although the alcohol Screening, Brief Intervention and Referral to Treatment (SBIRT) approach has shown promise as a low-cost, effective strategy for reducing alcohol use in civilians many of whom are risky drinkers but not yet dependent, it has not been adapted or tested in military health care settings for active duty personnel. This 2.5 year civilian-military collaborative study is highly responsive to exploring solutions to this emerging issue. The specific objectives for the overall project are given below.

Objective 1: Feasibility and Acceptability

* Determine how the SBIRT intervention can be integrated into standard military emergency department (ED) operations by conducting record review and observation of the ED.
* Develop and test the acceptability and usability (for both ED staff and potential participants) of the SBIRT approach by conducting focus groups with active duty personnel and garnering input from ED staff.
* Develop an implementation/operations protocol for delivering SBIRT in the ED.

Objective 2: Adaptation

* Apply a translational research approach to adapt SBIRT implementation in military settings and populations by using information from focus groups and input from ED staff.
* Adapt the content of the SBIRT intervention to be relevant for military personnel, including language and images for counseling and materials using information from focus groups and input from ED staff.

Objective 3: Pilot Trial

* Using a two group repeated measures design, assess the impact of SBIRT using standardized alcohol use measures to assess its potential for effectiveness with active duty military personnel in an ED setting. Specific methodologies include:
* Apply a randomization method in the ED to assign active duty participants to experimental condition.
* Implement the SBIRT intervention in the ED for those assigned to the intervention arm.
* Implement a process for obtaining follow-up data with this mobile population.
* Assess presumed mediators (e.g., readiness/motivation to change and self-efficacy) and moderators (e.g., PTSD status, gender) of alcohol misuse change.

ELIGIBILITY:
Inclusion Criteria:

* 18 or Older
* Active Duty
* Off Duty
* Telephone Number for Follow-up
* Healthy Enough to Participate
* Positive Screen for Risky Drinking

Exclusion Criteria:

* Under 18
* Non-Military
* On Duty
* Low Level Drinking

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 791 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Reed, PhD, Principal Investigator — SDSURF - Center for Alcohol & Drug Studies & Services; Gerard DeMers, DO, Principal Investigator — United States Naval Medical Center, San Diego
Locations (1):
- Naval Medical Center San Diego, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- SBIRT: Those assigned to the SBIRT intervention group will receive 1 of 3 tracks:
  1. Brief Intervention (BI) for At Risk Individuals (scores lower than 15) - Brief motivational intervention with feedback related to their use and change strategies.
  2. Brief Treatment (BT) for High Risk Individuals (scores of 16-19) - Brief Intervention on site and be offered 6 individual confidential sessions with a civilian Brief Treatment Counselor over the phone.
  3. Referral to Treatment (RT) for Severe Risk Individuals (scores of 20-40) - Brief Intervention on site and will be given a list of services where they may self-refer for further assessment and support.
  SBIRT: SBIRT is an "opportunistic" approach whereby patients are screened by Health Educators for their alcohol use, and then, taking advantage of a "teachable moment," are delivered a brief, motivational intervention matched to their level of risk.
Period: Overall Study
Arm/Group | Usual Care | SBIRT
Started | 403 | 388
Completed | 244 | 228
Not Completed | 159 | 160
Not completed — Lost to Follow-up | 146 | 142
Not completed — Withdrawal by Subject | 13 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | SBIRT | Total
Number analyzed (Participants) | 403 | 388 | 791
Age, Continuous [Mean (Standard Deviation); unit: Years] | 26.4 (6) | 26.3 (5.7) | 26.3 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 108 | 211
  Male | 300 | 280 | 580
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic/Latino | 85 | 64 | 149
  African-American | 74 | 71 | 145
  White | 215 | 214 | 429
  Asian/Hawaiian/Pacific Islander | 10 | 15 | 25
  American Indian/Alaskan Native | 4 | 2 | 6
  Other | 15 | 22 | 37
Region of Enrollment [Number; unit: participants]
  United States | 403 | 388 | 791
Self-Reported PTSD Diagnosis [Count of Participants; unit: Participants]
  Yes | 16 | 21 | 37
  No | 387 | 367 | 754
Marital Status [Count of Participants; unit: Participants]
  Single | 203 | 185 | 388
  Married/Co-habitating | 161 | 173 | 334
  Divorced/Separated/Widowed | 39 | 30 | 69
Education Level [Count of Participants; unit: Participants]
  High School Graduate/GED | 169 | 149 | 318
  Some College | 123 | 128 | 251
  2-Year College Degree (AA) | 52 | 43 | 95
  4-Year Degree (BA/BS) | 46 | 50 | 96
  Graduate Degree | 13 | 18 | 31
Service Branch [Count of Participants; unit: Participants]
  Navy | 336 | 320 | 656
  Marine Corps | 57 | 54 | 111
  Army/Air Force/Coast Guard | 9 | 14 | 23
  Missing | 1 | 0 | 1
Number of Combat Deployments (past 5-years) [Count of Participants; unit: Participants]
  None | 211 | 214 | 425
  1-2 | 173 | 148 | 321
  3 or more | 19 | 25 | 44
  Missing | 0 | 1 | 1
Alcohol Use Disorders Identification Test (AUDIT) Score [Mean (Standard Deviation); unit: units on a scale] — The AUDIT is the Alcohol Use Disorders identification test (Babor et al., 2001). The AUDIT is a screening assessment designed to help identify risky drinking. The AUDIT ranges from a score of 0 to 40 with higher values indicating riskier drinking.
  units on a scale | 7.7 (4.2) | 8.0 (5.1) | 7.7 (4.6)
Readiness to Change Drinking [Mean (Standard Deviation); unit: units on a scale] — A readiness to change alcohol use measure (ranging from 1 - not ready to change, to 4 - very ready) was assessed at baseline and follow-up for all participants. Because motivation and readiness to change are hallmark elements of the SBIRT approach and are thought to be integral to behavior change, these constructs will be measured to assess the degree to which they change in the two groups. Some individuals may not abstain or reduce their use over time, but there may be an improvement in their readiness to change.
  units on a scale | 1.95 (1.17) | 1.96 (1.15) | 1.96 (1.16)
Controlled Drinking Self-Efficacy Scale (CDSES) [Mean (Standard Deviation); unit: units on a scale] — The 20-item Controlled Drinking Self-Efficacy Scale (CDSES; Sitharthan et al., 2003), is a reliable, valid, easy-to-administer scale that assesses confidence to reduce overall consumption and frequency of drinking. Items range from 0% to 100% with higher scores indicating more confidence to engage in controlled drinking. Items for the CDSES will be combined and averaged to form a scaled score.
  units on a scale | 76.9 (15.3) | 78 (15) | 77.9 (15.2)

OUTCOME MEASURES:

1. Primary Outcome: Alcohol Use Disorders Identification Test (AUDIT) Total
Description: The primary outcome measure will come from the participant's total score on the AUDIT. Scores on the AUDIT range from 0 to 40 with higher numbers indicating greater problematic alcohol use. Mean AUDIT scores at follow-up will be compared between arms.
Time Frame: Baseline, Follow-up (Up to 7 months)
Population: Excludes low-risk participants defined as AUDIT <=7 at baseline. A total of 17 participants were excluded from the analysis.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Usual Care | SBIRT
Number analyzed (Participants) | 240 | 215
units on a scale | 5.91 (0.26) | 5.5 (0.27)
Statistical Analysis 1: Comparison: Usual Care vs SBIRT; Data were analyzed using a GLM repeated measures approach. A priori means comparisons tests (usual care vs. SBIRT intervention) with Bonferroni corrections were used to compare mean differences at follow-up; Test type: Other; p = 0.274, Repeated Measures--General Linear Model — A priori threshold for statistical significance was 0.05

2. Secondary Outcome: AUDIT-C or Drinkers Index
Description: The drinkers index consists of a summary of the first three AUDIT items which represents a combination of quantity, usual frequency, and frequency of heavy drinking. The AUDIT-C can range from 0 to 12 with 12 representing higher levels of drinking quantity and frequency.
Time Frame: Baseline, Follow-up (Up to 7 months)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Usual Care | SBIRT
Number analyzed (Participants) | 240 | 215
units on a scale | 4.41 (0.14) | 4.05 (0.15)
Statistical Analysis 1: Comparison: Usual Care vs SBIRT; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.083, Repeated Measures--General Linear Model

3. Secondary Outcome: Controlled Drinking Self-Efficacy Scale (CDSES)
Description: The 20-item Controlled Drinking Self-Efficacy Scale (CDSES), is a reliable, valid, easy-to-administer scale that assesses confidence to reduce overall consumption and frequency of drinking. Items range from 0% to 100% with 100% indicating more confidence to engage in controlled drinking. The CDSES was administered at both baseline and follow-up to assess changes in this presumed mediating attitude.
Time Frame: Baseline, Follow-up (Up to 7 months)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Usual Care | SBIRT
Number analyzed (Participants) | 240 | 215
units on a scale | 78.42 (1.01) | 81.67 (1.07)
Statistical Analysis 1: Comparison: Usual Care vs SBIRT; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.028, Repeated Measures--General Linear Model

4. Secondary Outcome: Readiness to Change Scale
Description: A readiness to change alcohol use measure (ranging from 1 - not ready to change, to 4 - very ready) was assessed at baseline and follow-up for all participants. Because motivation and readiness to change are hallmark elements of the SBIRT approach and are thought to be integral to behavior change, these constructs will be measured to assess the degree to which they change in the two groups. Some individuals may not abstain or reduce their use over time, but there may be an improvement in their readiness to change.
Time Frame: Baseline, Follow-up (Up to 7 months)
Population: Excludes low-risk participants defined as AUDIT <=7 at baseline. A total of 17 participants were excluded from the analysis as they were low-risk at baseline. Additionally, missing data on the Readiness to Change measure resulted in a total of 444 participants for this analysis. Six were missing from usual care and five were missing from SBIRT.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Usual Care | SBIRT
Number analyzed (Participants) | 234 | 210
units on a scale | 2.23 (0.08) | 2.19 (0.09)
Statistical Analysis 1: Comparison: Usual Care vs SBIRT; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.708, Repeated Measures--General Linear Model

5. Post Hoc Outcome: Alcohol Use Disorders Identification Test (AUDIT) Total (Analysis II)
Description: as for outcome 1
Time Frame: Baseline, Follow-up (Up to 7 months)
Population: For this study, at-risk drinking was defined as: AUDIT total >=8, under 21 drinker, any past year heavy episodic drinking (HED). Excludes at-risk participants defined as any amount of HED (AUDIT Question 3 > 0) or under 21 drinker at baseline. A total of 281 participants were excluded from this analysis (N = 190)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Usual Care | SBIRT
Number analyzed (Participants) | 100 | 90
units on a scale | 8.2 (0.47) | 7.31 (0.34)
Statistical Analysis 1: Comparison: Usual Care vs SBIRT; Data were analyzed using a GLM repeated measures approach. A priori means comparisons tets (usual care vs. SBIRT intervention) with Bonferroni corrections were used to compare mean differences at follow-up; Test type: Other; p = 0.197, Repeated Measures--General Linear Model — A priori threshold for statistical significance was 0.05

6. Post Hoc Outcome: AUDIT-C or Drinkers Index (Analysis II)
Description: as for outcome 2
Time Frame: Baseline, Follow-up (Up to 7 months)
Population: as for outcome 5
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Usual Care | SBIRT
Number analyzed (Participants) | 100 | 90
units on a scale | 5.42 (0.24) | 4.63 (0.25)
Statistical Analysis 1: Comparison: Usual Care vs SBIRT; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.023, Repeated Measures--General Linear Model — A priori threshold for statistical significance was 0.05

7. Post Hoc Outcome: Controlled Drinking Self-Efficacy Scale (CDSES) (Analysis II)
Description: as for outcome 3
Time Frame: Baseline, Follow-up (Up to 7 months)
Population: as for outcome 5
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Usual Care | SBIRT
Number analyzed (Participants) | 100 | 89
units on a scale | 70.45 (1.55) | 79.34 (1.65)
Statistical Analysis 1: Comparison: Usual Care vs SBIRT; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < 0.001, Repeated Measures--General Linear Model — A priori threshold for statistical significance was 0.05

8. Post Hoc Outcome: Readiness to Change Scale (Analysis II)
Description: as for outcome 4
Time Frame: Baseline, Follow-up (Up to 7 months)
Population: as for outcome 5
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Usual Care | SBIRT
Number analyzed (Participants) | 98 | 89
units on a scale | 2.29 (0.13) | 2.46 (0.14)
Statistical Analysis 1: Comparison: Usual Care vs SBIRT; Data were analyzed using a GLM repeated measures approach. A priori means comparison tests (usual care vs. SBIRT intervention) with Bonferroni corrections were used to compare means differences at follow-up; Test type: Other; p = 0.348, Repeated Measures--General Linear Model — A priori threshold for statistical significance was 0.05

9. Post Hoc Outcome: Alcohol Use Disorders Identification Test (AUDIT) Total (Analysis III--complete Cases)
Description: as for outcome 1
Time Frame: Baseline, Follow-up (Up to 7 months)
Population: Complete case analysis
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Usual Care | SBIRT
Number analyzed (Participants) | 244 | 227
units on a scale | 5.87 (0.25) | 5.48 (0.26)
Statistical Analysis 1: Comparison: Usual Care vs SBIRT; [analysis description as in outcome 8, analysis 1]; Test type: Other; p = 0.091, Repeated Measures GLM — A priori threshold for statistical significance was 0.05; Mean Difference (Final Values) = .345, Standard Error of Mean .203

10. Post Hoc Outcome: AUDIT-C or Drinkers Index (Analysis III Complete Cases)
Description: as for outcome 2
Time Frame: Baseline, Follow-up (Up to 7 months)
Population: Complete case analysis
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Usual Care | SBIRT
Number analyzed (Participants) | 244 | 227
units on a scale | 4.4 (.14) | 4.05 (.15)
Statistical Analysis 1: Comparison: Usual Care vs SBIRT; [analysis description as in outcome 8, analysis 1]; Test type: Other; p = .278, Repeated Measures GLM — A priori alpha set at 0.05; Mean Difference (Net) = .393, Standard Error of Mean .362

11. Post Hoc Outcome: Controlled Drinking Self-Efficacy Scale (CDSES) (Analysis III Complete Cases)
Description: as for outcome 3
Time Frame: Baseline, Follow-up (Up to 7 months)
Population: Complete case analysis
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Usual Care | SBIRT
Number analyzed (Participants) | 244 | 227
units on a scale | 78.66 (1.0) | 81.82 (1.04)
Statistical Analysis 1: Comparison: Usual Care vs SBIRT; [analysis description as in outcome 8, analysis 1]; Test type: Other; p = 0.029, Repeated Measures GLM — A priori alpha set at 0.05; Mean Difference (Net) = 3.163, Standard Error of Mean 1.44

12. Post Hoc Outcome: Readiness to Change Scale (Analysis III Complete Cases)
Description: as for outcome 4
Time Frame: Baseline, Follow-up (Up to 7 months)
Population: Complete case analysis
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Usual Care | SBIRT
Number analyzed (Participants) | 238 | 221
units on a scale | 2.21 (0.08) | 2.20 (0.09)
Statistical Analysis 1: Comparison: Usual Care vs SBIRT; [analysis description as in outcome 8, analysis 1]; Test type: Other; p = 0.897, Repeated Measures GLM — A priori alpha set at 0.05; Mean Difference (Net) = -0.015

13. Post Hoc Outcome: Alcohol Use Disorders Identification Test (AUDIT) Total (Analysis IV--Multiple Imputation and Intention to Treat Analysis)
Description: as for outcome 1
Time Frame: Baseline, Follow-up (Up to 7 months)
Population: Intent to treat analysis using multiple imputation; include all participants allocated to a condition at baseline (n = 791)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Usual Care | SBIRT
Number analyzed (Participants) | 403 | 388
units on a scale | 4.47 (0.16) | 4.15 (0.13)
Statistical Analysis 1: Comparison: Usual Care vs SBIRT; Linear mixed-effects models were used to analyze 5 pooled datasets derived from multiple imputation for intent to treat analyses; Test type: Other; p = 0.15, Linear mixed effects

14. Post Hoc Outcome: AUDIT-C or Drinkers Index (Analysis IV--Intent to Treat Analyses)
Description: as for outcome 2
Time Frame: Baseline, Follow-up (Up to 7 months)
Population: as for outcome 13
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Usual Care | SBIRT
Number analyzed (Participants) | 403 | 388
units on a scale | 5.95 (0.21) | 5.62 (0.23)
Statistical Analysis 1: Comparison: Usual Care vs SBIRT; [analysis description as in outcome 13, analysis 1]; Test type: Other; p = 0.20, Linear mixed effects — A priori alpha set at 0.05

15. Post Hoc Outcome: Controlled Drinking Self-Efficacy Scale (CDSES) (Analysis IV--Intent to Treat Analyses)
Description: as for outcome 3
Time Frame: Baseline, Follow-up (Up to 7 months)
Population: as for outcome 13
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Usual Care | SBIRT
Number analyzed (Participants) | 403 | 388
units on a scale | 78.42 (0.85) | 81.30 (1.05)
Statistical Analysis 1: Comparison: Usual Care vs SBIRT; [analysis description as in outcome 13, analysis 1]; Test type: Other; p = 0.38, Linear mixed effects — A priori alpha set at 0.05

16. Post Hoc Outcome: Readiness to Change Scale (Analysis IV--Multiple Imputation and Intention to Treat Analysis)
Description: as for outcome 4
Time Frame: Baseline, Follow-up (Up to 7 months)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Usual Care | SBIRT
Number analyzed (Participants) | 403 | 388
units on a scale | 2.22 (0.07) | 2.16 (0.07)
Statistical Analysis 1: Comparison: Usual Care vs SBIRT; [analysis description as in outcome 13, analysis 1]; Test type: Other — A priori alpha set at 0.05; p = 0.48, Linear mixed effects

17. Post Hoc Outcome: Alcohol Use Disorders Identification Test (AUDIT) Total (Analysis V--Multiple Imputation and Intention to Treat Analysis)
Description: as for outcome 1
Time Frame: Baseline, Follow-up (Up to 7 months)
Population: Intent to treat analysis using multiple imputation; includes participants scoring 8 or greater on the AUDIT at baseline.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Usual Care | SBIRT
Number analyzed (Participants) | 166 | 161
units on a scale | 5.38 (0.25) | 4.85 (0.20)
Statistical Analysis 1: Comparison: Usual Care vs SBIRT; [analysis description as in outcome 13, analysis 1]; Test type: Other — A priori alpha set at 0.05; p = 0.09, Linear mixed effects

18. Post Hoc Outcome: AUDIT-C or Drinkers Index (Analysis V--Intent to Treat Analyses)
Description: as for outcome 2
Time Frame: Baseline, Follow-up (Up to 7 months)
Population: Intent to treat analysis using multiple imputation; includes participants scoring 8 or greater on the AUDIT at baseline.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Usual Care | SBIRT
Number analyzed (Participants) | 166 | 161
units on a scale | 8.09 (0.39) | 7.64 (0.38)
Statistical Analysis 1: Comparison: Usual Care vs SBIRT; A priori alpha set at 0.05; Test type: Other; p = 0.08, Linear mixed effects

19. Post Hoc Outcome: Controlled Drinking Self-Efficacy Scale (CDSES) (Analysis V--Intent to Treat Analyses)
Description: as for outcome 3
Time Frame: Baseline, Follow-up (Up to 7 months)
Population: Intent to treat analysis using multiple imputation; includes participants scoring 8 or greater on the AUDIT at baseline.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Usual Care | SBIRT
Number analyzed (Participants) | 166 | 161
units on a scale | 72.18 (1.38) | 77.84 (1.55)
Statistical Analysis 1: Comparison: Usual Care vs SBIRT; A priori alpha set at 0.05; Test type: Other; p = 0.11, Linear mixed effects

20. Post Hoc Outcome: Readiness to Change Scale (Analysis V--Multiple Imputation and Intention to Treat Analysis)
Description: as for outcome 4
Time Frame: Baseline, Follow-up (Up to 7 months)
Population: Intent to treat analysis using multiple imputation; includes participants scoring 8 or greater on the AUDIT at baseline.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Usual Care | SBIRT
Number analyzed (Participants) | 166 | 161
units on a scale | 2.33 (0.10) | 2.35 (0.12)
Statistical Analysis 1: Comparison: Usual Care vs SBIRT; A priori alpha set at 0.05; Test type: Other; p = 0.84, Linear mixed effects

ADVERSE EVENTS:
Arm/Group | Usual Care | SBIRT
Serious Adverse Events (participants affected / at risk) | 0/244 | 0/228
Other Adverse Events (participants affected / at risk) | 0/244 | 0/228

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No